CLINICAL TRIAL: NCT02818127
Title: Assessment Of Total Coronary Circulation Time Using TIMI Frame Count Method In Patients Undergoing Coronary Angiography
Brief Title: Assessment Of Total Coronary Circulation Time Using TIMI Frame Count Method (TCCT-TIMI)
Acronym: TCCT-TIMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vascular and Molecular Cardiology Society (Other)
Collaborators: Private Yenisehir Hospital (Unknown); Private Gozde Hospital (Unknown); Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Vasmol002
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Angiography; Coronary Artery Disease; Coronary Artery Ectasia; Slow-Flow Phenomenon; Coronary Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Aneurysm; No-Reflow Phenomenon; Coronary Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- normal coronary artery (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- coronary slow flow (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- coronary artery ectasia (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- non-obstructive coronary artery disease (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- obstructive coronary artery disease (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: coronary angiography — Coronary angiography will be performed by transfemoral or transradial approach in all patients. In order to evaluate each coronary artery, at least four views from the left and two views from the right system will be taken.

SUMMARY:
The aim of this study is to evaluate and describe the total coronary circulation time (TCCT) by using TIMI frame count method in patients performed coronary angiography. TCCT is described as an angiographic index which is the sum of the frame count of coronary artery and venous system. This study also evaluates the relationship between the diseases in arterial system such as coronary artery ectasia, coronary slow flow, coronary artery disease and coronary venous pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom performed coronary angiography with a suspicion of coronary artery disease

Exclusion Criteria:

* History of cerebrovascular disease, chronic inflamatuar disease, malignity, chronic kidney and hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of total coronary circulation time by using TIMI frame count method | 1 day

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Gulhane Military Medical Academy, Ankara, Kecioren
  - Private Gozde Hospital, Malatya
  - Private Yenisehir Hospital, Mersin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] von Ludinghausen M. The venous drainage of the human myocardium. Adv Anat Embryol Cell Biol. 2003;168:I-VIII, 1-104. doi: 10.1007/978-3-642-55623-4. PMID 12645157
- [Background] Gibson CM, Cannon CP, Daley WL, Dodge JT Jr, Alexander B Jr, Marble SJ, McCabe CH, Raymond L, Fortin T, Poole WK, Braunwald E. TIMI frame count: a quantitative method of assessing coronary artery flow. Circulation. 1996 Mar 1;93(5):879-88. doi: 10.1161/01.cir.93.5.879. PMID 8598078